CLINICAL TRIAL: NCT04547114
Title: Breath Analysis for SARS-CoV-2 in Infected and Healthy Subjects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Klinikum Bayreuth GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: IMS COVID-19
Record Dates: First submitted 2020-09-11; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SARS-CoV-2- infected: Detection of SARS-CoV-2 RNA by PCR in nasopharyngeal/oropharyngeal swabs
  Interventions: Diagnostic Test: Multicapillary column coupled ion mobility spectrometry
- non infected: Lack of detection of SARS-CoV-2 RNA by PCR in nasopharyngeal/oropharyngeal swabs
  Interventions: Diagnostic Test: Multicapillary column coupled ion mobility spectrometry

INTERVENTIONS:
Diagnostic Test: Multicapillary column coupled ion mobility spectrometry — sampling of nasal air via a foam cuffed oxygen catheter

SUMMARY:
Recently published studies could demonstrate that detection of specific biomarkers in breath could be applied for the diagnosis of SARS-CoV-2.

DETAILED DESCRIPTION:
In this study we want to address the sensitivity and specificity of breath analysis by MCC-IMS in the context of SARS-CoV-2 detection from PCR- proven infected and non-infected subjects.

Therefore nasal breath will be aspirated for 10 seconds during normal respiration by a foam cuffed oxygen catheter connected via a 0.22μm filter and a line into the MCC-IMS and directly analyzed without any pre-analytic procedures.

The during the proof-of-concept study derived significant peaks for volatile organic compounds will be used for discrimination in a point-of-care approach.

ELIGIBILITY:
Inclusion Criteria:

hospital admission staff members

Exclusion Criteria:

too sick to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult subjects of all genders and ages
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-09-14 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
correct classification of SARS-CoV-2 infected and not infected subjects | 6 months
  correct classification of SARS-CoV-2 infected and not infected subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Bayreuth/ Bayreuth General Hospital, Bayreuth, Germany

IPD SHARING:
Plan to Share IPD: No